CLINICAL TRIAL: NCT06477107
Title: Augmenting Cerebral Perfusion With Transcranial Direct Current Stimulation (tDCS) in Chronic Hypoperfusion States
Brief Title: A Study of Cerebral Perfusion With tDCS in Chronic Hypoperfusion
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Zafer Keser, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 24-001186
Record Dates: First submitted 2024-06-06; First posted 2024-06-27 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Moyamoya Syndrome; Moyamoya Disease; Atheroscleroses, Cerebral
MeSH Terms: conditions — Moyamoya Disease; Intracranial Arteriosclerosis

STUDY DESIGN:
Intervention Model Description: For the Phase I portion of the study subjects the order of the stimulation (active vs sham stimulation) in a single session will be randomized and counterbalanced across subjects.
  For the Phase II portion of the study a cross-over design will be used and the subjects will be randomly assigned either to active or sham tDCS first, then they will cross over to the other treatment arm after 4-week period of washout.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (6):
- Phase I - Health Volunteer Group: Active Stimulation, Then Sham Stimulation (Experimental): Healthy subjects will receive 20 minutes of 2 mA tDCS concurrently with MRI cerebral blood flow (CBF) imaging immediately followed by no stimulation and CBF imaging. Next, subjects will receive sham stimulation concurrently with CBF imaging immediately followed by no stimulation and CBF imaging.
  Interventions: Device: Soterix® 4x1HD-TDCS
- Phase I - Health Volunteer Group: Sham Stimulation, Then Active Stimulation (Experimental): Healthy subjects will receive sham stimulation concurrently with MRI CBF imaging immediately followed by no stimulation and CBF imaging. Next, subjects will receive 20 minutes of 2 mA tDCS concurrently with CBF imaging immediately followed by no stimulation and CBF imaging.
  Interventions: Device: Soterix® 4x1HD-TDCS
- Phase I Disease Group: Active Stimulation, Then Sham Stimulation (Experimental): Subject diagnosed with Moyamoya disease or severe extracranial atherosclerotic disease will receive 20 minutes of 2 mA tDCS concurrently with MRI cerebral blood flow (CBF) imaging immediately followed by no stimulation and CBF imaging. Next, subjects will receive sham stimulation concurrently with CBF imaging immediately followed by no stimulation and CBF imaging.
  Interventions: Device: Soterix® 4x1HD-TDCS
- Phase I Disease Group: Sham Stimulation, Then Active Stimulation (Experimental): Subject diagnosed with Moyamoya disease or severe extracranial atherosclerotic disease will receive sham stimulation concurrently with MRI CBF imaging immediately followed by no stimulation and CBF imaging. Next, subjects will receive 20 minutes of 2 mA tDCS concurrently with CBF imaging immediately followed by no stimulation and CBF imaging.
  Interventions: Device: Soterix® 4x1HD-TDCS
- Phase II Active Stimulation, Then Sham Stimulation (Experimental): Subjects first receive active tDCS plus cognitive training every weekday for 10 days. After washout period of 4 weeks, they will perform at-home sham tDCS plus cognitive training every weekday for 10 days.
  Interventions: Device: Soterix® 1x1 tDCS; Behavioral: Cognitive training program
- Phase II Sham Stimulation, Then Active Stimulation (Experimental): Subjects first receive sham tDCS plus cognitive training daily for 10 days. After a washout period of 4 weeks, they will perform at-home active tDCS plus cognitive training daily for 10 days.
  Interventions: Device: Soterix® 1x1 tDCS; Behavioral: Cognitive training program

INTERVENTIONS:
Device: Soterix® 4x1HD-TDCS — Is intended for inducing cortical neuromodulation for research and treatment purposes.
  Arms: Phase I - Health Volunteer Group: Active Stimulation, Then Sham Stimulation; Phase I - Health Volunteer Group: Sham Stimulation, Then Active Stimulation; Phase I Disease Group: Active Stimulation, Then Sham Stimulation; Phase I Disease Group: Sham Stimulation, Then Active Stimulation
Device: Soterix® 1x1 tDCS — At-home remotely supervised transcranial direct current stimulation (tDCS) at an intensity of 2 mA for 20 minutes per session, with slow ramp-up and automatic turn off once it reaches the maximal intensity.
  Arms: Phase II Active Stimulation, Then Sham Stimulation; Phase II Sham Stimulation, Then Active Stimulation
Behavioral: Cognitive training program — Computerized cognitive therapy for 45 minutes per day that starts at the same time with stimulation
  Arms: Phase II Active Stimulation, Then Sham Stimulation; Phase II Sham Stimulation, Then Active Stimulation

SUMMARY:
This study is being done to examine whether transcranial direct current stimulation (tDCS) will increase cerebral blood flow which may provide a clinical benefit such as improving cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Vasculopathy leading to imaging evidence of hypoperfusion
* Cognitive impairment

Exclusion Criteria:

* Pregnancy
* Contraindication to MRI or tDCS including metallic implanted objects.
* Medical instability or inability to cooperate during the study as assessed by the treating physician to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Changes in cerebral blood flow | Phase 1 Day 0 and Phase 2 Day 0, 14, 44, and 58
  Cerebral blood flow imaging assessed by MRI to measure blood flow through the blood vessels reported in millimeters of mercury (mmHg)

SECONDARY OUTCOMES:
Change in cognitive impairment | Phase 2 Days 0, 14±3, 44±7, and 58±14, 72±14
  Assessed using the Montreal Cognitive Assessment (MoCA), which is a 30-item questionnaire that includes tests of orientation, attention, memory, language and visual-spatial skills. Possible total scores range from 0 to 30, with higher scores indicating higher cognitive function. A final total score of 26 and above is consider normal.
Change in Fatigue Severity Scale (FFS) | Phase 2 Days 0, 14±3, 44±7, and 58±14, 72±14
  Assessed using the Fatigue Severity Scale (FFS) 9-item questionnaire that contains statements that rate fatigue symptoms on a scale of 1 to 7 where a low value (e.g., 1) indicates strong disagreement with the statement and a high value (e.g., 7) indicates strong agreement. Possible total scores range from 9 to 63, with higher scores indicating greater fatigue severity.
Change in Visual Analogue Scale to Evaluate Fatigue Severity (VAS-F) | Phase I Day 0, Phase 2 Days 0, 14±3, 44±7, and 58±14, 72±14
  Assessed using the Visual Analogue Scale to Evaluate Fatigue Severity (VAS-F) 18-item questionnaire that rates how a subject is currently feeling in regards to fatigue symptoms on a scale of 0 to 10 where a low value (e.g., 0) indicates "not at all/no effort at all" and a high value (e.g., 10) indicates "extremely/tremendous chore". Possible total scores range from 0 to 180, with higher scores indicating greater fatigue severity.
Change in Stroke Specific Quality of Life (SS-QOL) | Phase 2 Days 0, 14±3, 44±7, and 58±14, 72±14
  Assessed using the Stroke Specific Quality of Life (SS-QOL) 49-item questionnaire assessing quality of life with regards to energy, family roles, language, mobility, mood, personality, self-care, social roles, thinking, upper extremity function, vision, and work/productivity on a scale of 1 to 5 where a low value (e.g., 1) indicates "total help/couldn't do it at all/strongly agree" and a high value (e.g., 5) indicates "no help needed/no trouble at all/strongly disagree". Possible total scores range from 49 to 245, with higher scores indicating better quality of life.
Change in depression severity | Phase 2 Days 0, 14±3, 44±7, and 58±14, 72±14
  Assessed using the Patient Health Questionnaire 9-item (PHQ-9) scale to assess severity of depression. Scoring is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." Total score for the nine items ranges from 0 to 27 where 0 is no depression, 1-4 is minimal depression, 5-9 is mild depression, 10-14 is moderate depression, and 15-19 is moderately severe depression and 20-27 severe depression.
Change in sleepiness | Phase 2 Days 0, 14±3, 44±7, and 58±14, 72±14
  Assessed using the Epworth sleepiness scale (ESS) 8-item questionnaire that measures daytime sleepiness in participants. Possible scores range from 0-24, with higher scores indicating a higher average sleep propensity in daily life, and a worse outcome.
Change in trail making test | Phase 2 Days 0, 14±3, 44±7, and 58±14, 72±14
  The Trail Making Test is a two part assessment of cognitive functions, principally attention and working memory. Subjects connect a set of 25 dots as quickly as possible, connect 13 dots labeled alphabetically, and 12 dots that are numbered in an alternating pattern as quickly as possible without lifting the pen. Results are reported as the number of seconds required to complete the task with higher scores indicating greater impairment.
Change in memory task | Phase 2 Days 0, 14±3, 44±7, and 58±14, 72±14
  Assessed using the Consortium to Establish a Registry for Alzheimer's Disease (CERAD) wordlist memory test (WLT). This is a memory task for assessing word list recall. A list of 10 words are read 3 times and subjects are asked to recall the list of words. The more words recalled indicates less cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Zafer Keser, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No